CLINICAL TRIAL: NCT06309706
Title: A Retrospective Cone Beam Computed Tomography Study of The Lateral Wall Bony Window
Status: Completed | Type: Observational
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: JXHU
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Lateral Wall Thickness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cross-sectional: To analyze the maxillary sinus anatomy over edentulous ridges in the bilateral posterior maxillary area in Chinese patients using cone-beam computed tomography (CBCT).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Just observation

SUMMARY:
Three experienced observers were asked to screen all the CBCT images from the Stomatology Hospital,Zhejiang University School of Medicine, between September 1, 2019 and December 31, 2019, and counted 1000 maxillary sinus CBCT images that met the criteria. Later, 1000 CBCT images were further measured and analyzed, and indicators such as maxillary sinus buccal wall thickness, morphology, whether there is blood vessel or not, whether there is bone septa or not were counted. The variation rules and related factors were summarized by SPSS analysis.

ELIGIBILITY:
Inclusion Criteria:

* Images were included if the following criteria were met: (1) patients were 18 years or older, (2) presence of teeth adjacent to or opposing the edentulous area allowing the location of the edentulous ridges corresponding to the tooth site to be identified, (3) presence of maxillary dentition defect in any tooth positon of the second premolar, the first molar or the second molar, (4) the maxillary sinus to be measured was visible from its floor to at least 15 mm high.

Exclusion Criteria:

* Images were excluded if any of the following criteria were met: (1) images were unclear or incomplete due to scattering or other reasons, (2) pristine maxillary posterior extraction sites after less than 3 months of healing and the tooth extraction sockets could be obviously identified, (3) the maxillary sinus had been grafted for implant-supported prosthesis, (4) implants or other prosthetic devices were present in maxillary posterior edentulous position, (5) orthodontic brackets and wires in images were present; (6) the location of the edentulous sites could not be determined, (7) sinus pathology was present that made the measurement impossible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: edentulous ridges in the bilateral posterior maxillary area in Chinese patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Lateral wall thickness | 2019-09-01~2019-12-31
  The thickness of the maxillary sinus lateral wall

CONTACTS AND LOCATIONS:
Locations (1):
- Stomatology Hospital, School of Stomatology, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Starch-Jensen T, Jensen JD. Maxillary Sinus Floor Augmentation: a Review of Selected Treatment Modalities. J Oral Maxillofac Res. 2017 Sep 30;8(3):e3. doi: 10.5037/jomr.2017.8303. eCollection 2017 Jul-Sep. PMID 29142655
- [Background] Monje A, Urban IA, Miron RJ, Caballe-Serrano J, Buser D, Wang HL. Morphologic Patterns of the Atrophic Posterior Maxilla and Clinical Implications for Bone Regenerative Therapy. Int J Periodontics Restorative Dent. 2017 Sep/Oct;37(5):e279-e289. doi: 10.11607/prd.3228. PMID 28817142